CLINICAL TRIAL: NCT01394484
Title: Milk and Yogurt vs. Calcium and Vitamin D Supplements for Bone Health of Women
Brief Title: Dairy Foods Compared to Dietary Supplements and Bone Health
Acronym: FL-83
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: WHNRC 201018566-1
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Osteoporosis; Bone Loss; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Four servings of dairy foods per day for 42 days, followed by washout for 42 days, followed by dietary supplements for 42 days
  Interventions: Other: Intervention I; Dietary Supplement: Intervention II
- Arm 2 (Experimental): Dietary Supplements for 42 days, followed by washout for 42 days, followed by 4 servings of dairy foods for 42 days.
  Interventions: Other: Intervention I; Dietary Supplement: Intervention II

INTERVENTIONS:
Other: Intervention I — Four servings of dairy foods (milk and yogurt) per day for 42 days.
Dietary Supplement: Intervention II — 1200 mg of supplemental calcium and 400 IU of vitamin D3 for 42 days

SUMMARY:
Does the consumption of dairy foods reduce the rate of bone loss in older women more than calcium and vitamin D supplements.

DETAILED DESCRIPTION:
Research indicates that bone health is dependent on multiple nutrients, not just calcium and vitamin D, leading to the conclusion that calcium from sources that include other bone enhancing nutrients may be more effective in maintaining bone integrity than calcium and vitamin D supplements. Several studies have examined the effects of calcium intake from dairy foods on different indicators of bone health. Reducing the rate of bone loss in postmenopausal women can reduce the risk of osteoporosis related fractures. Therefore we propose to study the effectiveness of 4 servings of milk and yogurt per day for 42 days compared to calcium and vitamin D supplements for 42 days to reduce calcium loss from the skeleton in post menopausal women. Postmenopausal women, approximately 50-65 years of age, will be studied. Each volunteer will receive both interventions in a cross-over design, in random order, separated by a 42 day washout period.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 24 months since last menses
* No hormone therapy in the past 12 months
* Weight stable for the past 3 months
* Bone density T score -1.7 to 0.0
* No more than two dairy servings per day
* No history of inflammatory disorders
* No history of non-traumatic bone fracture
* No supplement use or willing to discontinue
* No lactose intolerance
* Willing to consume milk and yogurt

Exclusion Criteria:

* Less than 24 months since last menses
* Use of hormone therapy in past yr
* > 5 pound weight change in past 3 months
* Osteoporosis
* Regular >2 servings/d of dairy
* Auto-immune/inflammatory disorders
* History of non-traumatic bone fracture
* Unwilling to discontinue supplements
* Lactose intolerance
* Unwilling to eat yogurt or drink milk

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Ratio of 41Ca/40Ca excreted in urine | Days 0, 90, 120, 150, 180, 187, 194, 201, 208, 215, 222, 229, 236, 243, 250, 257, 264,271, 278, 285, 292, 299, and 306 of the study
  Subjects will be asked to collect 24 hour urine samples to establish each individual's kinetic profile of Ca excretion and to measure the effectiveness of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Van Loan, PhD, Principal Investigator — WHNRC, ARS, University of California Davis; Marjorie Garrod, Ph.D., Study Director — USDA, ARS, WHNRC
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States